CLINICAL TRIAL: NCT06079138
Title: Tele-rehabilitation Using Transcranial Direct Current Stimulation Combined with Exercise in People with Spinal Cord Injury
Brief Title: Tele-rehabilitation Using TDCS Combined with Exercise in People with Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2023/119.0504
Record Dates: First submitted 2023-06-25; First posted 2023-10-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injury; Incomplete Spinal Cord Injury
Keywords: rehabilitation; home-based exercise; tDCS; SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The participants will be divided into 2 groups. Intervention group will receive active tDCS with intensity 2 mA and control group will receive sham tDCS.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS and telerehabilitation exercise program (Experimental): Participants will receive active tDCS with an intensity 2 mA for 20 minutes and a telerehabilitation exercise program for 50 minutes. The program will be implemented over 12 sessions, occurring three times a week for four weeks).
  Interventions: Device: Transcranial direct current stimulation (Active); Other: Telerehabilitation exercise
- Sham tDCS and Telerehabilitation exercise (Sham Comparator): Participants will receive sham tDCS for 20 minutes. The program will be implemented over 12 sessions, occurring three times a week for four weeks.
  Interventions: Device: Transcranial direct current stimulation (Sham); Other: Telerehabilitation exercise

INTERVENTIONS:
Device: Transcranial direct current stimulation (Active) — Participants will sit comfortably during the stimulation, and the scalp will be cleaned with alcohol beforehand. The Ybrain MINDD STIM current stimulator will be used with saline-soaked sponge-pad electrodes (35 cm2 in size). Electrode placement will follow the 10-20 EEG system, with the active (anodal) electrode (A) positioned at the vertex (Cz) on the more affected side and the reference (cathodal) electrode (C) placed over the supraorbital region on the less affected side. The electrodes will be attached to a cap before application.
  In the experimental group, participants will receive real tDCS at 2.0 mA for 20 minutes, with a 30-second ramp-up and ramp-down period.
  Other Names: tDCS (Active)
  Arms: Active tDCS and telerehabilitation exercise program
Device: Transcranial direct current stimulation (Sham) — Participants will sit comfortably during the stimulation, and the scalp will be cleaned with alcohol beforehand. The Ybrain MINDD STIM current stimulator will be used with saline-soaked sponge-pad electrodes (35 cm2 in size). Electrode placement will follow the 10-20 EEG system, with the active (anodal) electrode (A) positioned at the vertex (Cz) on the more affected side and the reference (cathodal) electrode (C) placed over the supraorbital region on the less affected side. The electrodes will be attached to a cap before application. The sham group will receive sham tDCS, where the current will only be delivered for the first 30 seconds and automatically stopped, while the electrodes remain in place for 20 minutes.
  Other Names: tDCS (Sham)
  Arms: Sham tDCS and Telerehabilitation exercise
Other: Telerehabilitation exercise — Telerehabilitation exercise will be provided via tele-conference meeting program. The program will consist of 3 parts. First part, there will be a limb exercise program for 20 minutes to prepare the joint range of motion and muscles. Second part, participants will receive functional balance training for 15 minutes to promote their postural balance during changing positions and static positions. Each exercise will perform 10 repetitions for each set and perform 3 sets. After 2-week of intervention, the set will be progressed to 4 sets. Final part, participants will receive 20 minutes of functional training of wheelchair/bed transferring exercise. Each wheelchair and bed transfer exercise will perform 10 repetitions for each completely transfer and perform 3 sets. After 2-week of intervention, the set will be progressed to 4 sets. After finishing all the programs, they will be asked to cool down by doing breathing exercises with torso stretching for 5 minutes.

SUMMARY:
This study aims to explore the effect of trans cranial direct current stimulation (tDCS) combined with self-exercise at home for 1 month training (3 sessions/week, for 4 weeks). The outcome assessment including motor function, functional activity, spasticity through neurological assessment (H reflex latency and H/M amplitude ratio) and quality of life will be assessed before, after the intervention and at 1- month follow-up. Participant will communicate with physical therapist via video online platform for every sessions (12 sessions).

DETAILED DESCRIPTION:
Spinal cord injury (SCI) can cause paralysis and functional disability, resulting in changes in strength and sensation. Rehabilitation is important for regaining independence, but short hospital stays and limited access to specialized clinics pose challenges. Telerehabilitation offers a solution by providing remote rehabilitation services.

Physical exercise and functional training are important for improving functional activity and endurance after SCI. Telerehabilitation has shown significant improvements in functional activity. However, the most effective gains occur within the first year after the injury, and rehabilitation training alone may not achieve full recovery. Impairments below the injury level can lead to changes in brain organization. Combining training with a top-down approach may promote motor recovery after SCI.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique used in neurorehabilitation. It can modulate neural activity in the primary motor cortex at both cortical and spinal levels and induce synaptic plasticity. Studies have shown that adjusting the intensity or duration of tDCS can enhance its effectiveness, with anodal stimulation increasing cortical excitability and cathodal stimulation decreasing it. Home-based tDCS is a safe, accessible, and convenient alternative to hospital-based tDCS. Previous research has suggested a positive trend for combining anodal tDCS with rehabilitation training in individuals with incomplete spinal cord injury. Strong arm endurance is crucial for individuals with complete SCI who require independent transfers and wheelchair use. Studies in healthy adults have demonstrated that tDCS combined with exercise can improve upper arm endurance. However, there is currently no research on the effects of tDCS combined with rehabilitation in improving functional skills for individuals with complete SCI, especially when applied through home-based tDCS with telerehabilitation.

In the early stages of spinal shock following a severe spinal cord injury (SCI), the H-reflex, a reflex measure of spinal cord excitability, is typically absent or significantly reduced below the injury site. The degree and duration of this reflex suppression indicate the severity of the injury. This loss of reflex activity is thought to result from decreased excitability of motoneurons due to the sudden loss of input from the brain. However, the H-reflex gradually starts to recover after the initial spinal shock phase. In patients with chronic complete spinal cord lesions, an increased H-reflex amplitude in the soleus muscle suggests heightened central synaptic excitability, which may contribute to the development of hyperreflexia after SCI. Recent research has shown that anodal tDCS can decrease the H/M ratio (the ratio of H-reflex to M-response) and H-reflex latency, leading to improved spasticity in patients with neurological conditions.

This study aims to investigate the impact of combining tDCS with self-exercise at home over a one-month training period. The training will involve three sessions per week for four weeks. The assessment will include measures of motor function, functional activity, spasticity (evaluated through neurological assessment of H-reflex latency and H/M amplitude ratio), and quality of life. The participants will interact with a physical therapist through a video online platform for each of the 12 sessions. Assessments will be conducted before and after the intervention, as well as at a one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with any level of SCI with age between 18-70 years.
* Onset of injury between 1-30 month.
* Must have electronic devices such as mobile phones or tablets or computers that can connect to the internet.

Exclusion Criteria:

* Receiving other NIBS and alternative medicine e.g. TMS, acupuncture.
* Having unstable cardiopulmonary disease e.g. unstable angina, uncontrolled atrial or ventricular arrythmias.
* Having uncontrolled conditions e.g. uncontrolled hypertension, uncontrolled diabetes.
* Having a history of other neurological diseases e.g. stroke.
* Having contra-indication to use tDCS (30) which are

  1. Having intracranial metal implantation, cochlear implant, or cardiac pacemaker.
  2. Having an open wound or wound infection on the scalp.
  3. Having a history of brain surgery.
  4. Having a history of epilepsy.

Ages: 18 Months to 70 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline: ASIA impairment scale | Baseline, post-intervention day 30, and 1-month after post-intervention
  The American spinal injury association is a universal classification tool for spinal cord injuries based on a standardized sensory and motor assessment, to determine the Sensory Level and Motor Level for each side of the body (Right and Left), the single Neurological Level of Injury (NLI) and whether the injury is Complete or Incomplete. For the Key Sensory point that related to the dermatomes C2 - S5. They are tested bilaterally using Light Touch (LT) (tested by cotton tip) and Pin-Prick (PP) [sharp-dull discrimination]. For motor examination, key motor function of the myotomes C5 - T1 and L2 - S1 are tested bilaterally.

SECONDARY OUTCOMES:
Change from baseline: the soleus H-reflex | Baseline, post-intervention day 30, and 1-month after post-intervention
  The soleus H-reflex is a monosynaptic response that is reliably elicited in the lower limb by stimulating the posterior tibial nerve (PTN) in the popliteal fossa. The H-reflex is evoked in the soleus muscle by percutaneous PTN stimulation with a 1 ms duration stimulus delivered at 0.33 Hz. Surface electrodes are used to record the H-reflex and motor (M) response from the soleus muscle. The M response represents direct motor activation, while the H-reflex appears later. The latency of the M response is 5-10 msec, while the H-reflex latency is 25-35 msec. Expressing the H-reflex as a percentage of the maximum M response (Mmax) allows for comparisons between individuals. The H-reflex response (Hmax) and Mmax will be recorded to calculate the H-reflex latency and H/M amplitude ratio.
Change from baseline: Modified Ashworth scale | Baseline, post-intervention day 30, and 1-month after post-intervention
  A clinical tool used to measure the increase of muscle tone.
Change from baseline: Upper limb muscle strength | Baseline, post-intervention day 30, 1-month after post-intervention
  This test will be used for assessing the improvement of upper limb muscle strength including shoulder flexor, shoulder abductor, shoulder extensor shoulder adductor, elbow flexor, wrist extensor, elbow extensor, and wrist flexor on both sides. The muscle strength will be assessed by using hand-held dynamometer (Lafayette Electronic Hand-held Dynamometer). This test had good reliability for testing in SCI. The participants will be asked to exert force against the dynamometer over a period second while the assessor will hold the dynamometer steady against their effort. The peak force (Newton) will be chosen for an outcome.
Change from baseline: Spinal cord independence measure III (SCIM III) | Baseline, post-intervention day 30, 1-month after post-intervention
  The Spinal Cord Independence Measure (SCIM) is a scale for the assessment of achievements of daily function of patients with spinal cord lesions (SCLs). The third version (SCIM III) contains 19 tasks organized in 3 subscales: self-care, respiration and sphincter management, and mobility. This study will assess only 2 subscales of self-care and mobility.
Change from baseline: Transfer assessment instrument (TAI) | Baseline, post-intervention day 30, 1-month after post-intervention
  The TAI evaluates wheelchair preparation, body setup, and flight phases of the transfer. It has good face, content, and construct validity for community-dwelling mobility device users. Each of the items in the TAI is scored "yes" (1 point), "no" (0 points), or "not applicable" (item not included in scoring), resulting in a minimum score of 0 and a maximum score of 10.
Change from baseline: Quality of life measure | Baseline, post-intervention day 30, 1-month after intervention
  The participants' QOL will also be evaluated by using the WHOQOL-BREF-Thai questionnaire that can be assessed by self-report. In situations that the participants cannot read, the assessor will read for them, and they will have to choose the answer by themselves. The WHOQOL-BREF questionnaire has two types of questions: perceived objective and self-report subjective, and it includes four components of well-being: physical, psychological, social, and environmental. Each item is scored from 1-5. This Thai version has a good internal consistency with Cronbach's alpha 0.84. The higher score indicates better QOL.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No